CLINICAL TRIAL: NCT06689696
Title: Pivotal Clinical Study to Evaluate the Smartlens miLens Measurement Performance and Safety Over a 24-hour Wear Period
Brief Title: 24-hour Wear Performance and Safety Study of Smartlens miLens Contact Lens for IOP Monitoring
Status: Recruiting | Type: Observational
Sponsor: Smartlens, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: miLens-002
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Glaucoma; GLAUCOMA 1, OPEN ANGLE, D (Disorder); Ocular Hypertension; Ocular Hypertension (OH); Ocular Hypertension Glaucoma; IOP; Intraocular Pressure; Glaucoma Open-Angle; Glaucoma and Ocular Hypertension; Glaucoma Patients and Healthy Controls; Normal Tension Glaucoma (NTG)
Keywords: IOP monitoring; Glaucoma; Contact lens for Glaucoma; Contact lens for IOP monitoring; IOP; Smart contact lens; POAG; Ocular Hypertension; Normal tension Glaucoma; IOP fluctuation
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- POAG: primary open angle glaucoma (POAG) including normal tension glaucoma
  Interventions: Device: miLens system
- POAG suspect: status as POAG suspect including ocular hypertension (OHTN)
  Interventions: Device: miLens system
- Healthy: no prior diagnosis of POAG/POAG suspect
  Interventions: Device: miLens system

INTERVENTIONS:
Device: miLens system — The miLens system consists of the miLens contact lens made of soft, biocompatible materials, the miLens imaging system, and miLens analysis software.

SUMMARY:
The goal of this clinical trial is to learn if a new contact lens device can record patterns in eye pressure for 24 hours in adults with glaucoma and in healthy participants.

The main questions it aims to answer are:

* Is the contact lens device able to detect patterns in eye pressure that happens naturally between nighttime and daytime?
* Are the contact lens recording patterns similar when repeated one week later?
* What eye problems do participants have when wearing contact lens for up to 24 hours?

Researchers will compare if the recordings detected by the contact lens over 24 hours are similar to the patterns measured by an eye pressure measuring instrument used in a doctor's office.

Participants will

* Wear contact lens in one eye for up to 24 hours
* Take recordings in that eye with smartphone camera every 15 minutes when awake
* For those participants who are able to stay overnight at a hotel for the trial, researchers will measure the eye pressure in the other eye every 1 to 2 hours when awake with an eye pressure measuring instrument.

DETAILED DESCRIPTION:
This study will enroll healthy participants and those with primary open-angle glaucoma or ocular hypertension from a minimum of two and up to 10 research sites in US.

All participants will be informed about the study and its potential risks and required to provide written informed consent prior to undergoing study-related procedures. Participants will be screened for eligibility. The study will be conducted in a 24-hour session in eligible subjects, preferably at a hotel or similar location that allows overnight stay. For subjects who complete the first session at a hotel and are able to return in a week, the study will be repeated in another 24-hour session.

At the beginning of the 24-hour session, the study staff will place the miLens in the study eye. The study eye is designated as the eye with higher intraocular pressure (IOP) or randomly selected if IOP is equal. Participants will be asked to capture miLens measurements using smartphone camera. The miLens smartphone app will auto-adjust zoom and capture image, which will be automatically sent to the cloud-based image processing software. The participants will be asked to capture miLens images every 15 minutes over 24 hours, except during sleep time between 10:30 pm and 5:30 am.

The study staff will also measure IOP in the other eye using a tonometer every 1-2 hours. In addition, participants will be asked to rate comfort on a numerical scale to assess tolerability to lens wear. Safety is assessed by biomicroscopy examination and by measuring vision and refraction before and after the session.

The 24-hour session is repeated after 6-8 days, starting at around the same time as the first session, in the same study eye.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥22 to ≤80 years of age
2. Subjects with:

   * prior diagnosis of POAG in at least one eye, including normal tension glaucoma or prior diagnosis of POAG suspect including OHTN in at least one eye for whom no evidence or suspicion of structural or functional glaucomatous damage exists

     * Diagnosis of POAG from medical records characterized by open angles and (1) optic nerve cupping consistent with glaucoma, with diffuse or focal thinning of neuroretinal rim or nerve fiber layer defects or a difference in cup/disc ratio > 0.2, not explained by anisometropia or other non-glaucomatous causes (2) visual field defects consistent with optic nerve cupping, with glaucomatous hemifield test outside normal limits or a pattern standard deviation (PSD) worse than 5th percentile (P<0.05) by Standard Automated Perimetry, or VF defects with Goldmann visual field test consistent with glaucomatous nerve fiber layer loss including paracentral scotoma, nasal step or arcuate defects
     * Diagnosis of POAG suspect from medical records established by open angles and IOP ≥22 mmHg (OHTN) OR abnormal appearing optic disc appearance OR glaucomatous visual field defects
   * no prior history of POAG/OHTN in either eye
3. In subjects with no history of POAG/OHTN, GAT IOP difference between eyes must be ≤ 2 mmHg, with IOP no less than 10 mmHg in both eyes and no greater than 21 mmHg in both eyes.
4. Mean keratometry value is between 7.5 mm and 8.2 mm in at least one eye (the miLens eye)
5. GEN4 miLens contact lens fitting on the subject's eye is acceptable by a slit lamp exam at Day 0 (measurement study visit)
6. Subjects with ability to discontinue habitual IOP-lowering medications, if any, in both eyes on Day 0 visit until the end of the 24-hour wear period (and if applicable, similarly for the Week 1 visit) (No preservative-free topical glaucoma medications will be allowed for the duration of the study)
7. Able to understand, sign and complete the informed consent and available to complete the minimum set of self-acquired smartphone images over the 24-hour contact lens wear period, preferably at an assigned site and likely available for a repeat session after a week

Exclusion Criteria:

1. BCVA worse than 20/200 in either eye
2. Greater than 6 diopters spherical equivalent in either eye
3. Greater than 3 diopters of keratometric cylinder in either eye
4. Central corneal thickness greater than 0.60 mm or less than 0.50 mm in either eye (per GAT study guidelines in ANSI Z80.10)
5. Known history of difficulty in obtaining Goldmann IOP measurements or any factors that might contribute to inaccurate Goldmann IOP measurements (e.g. lid squeezing or tremor)
6. Subjects who have had ocular surgery within the last 6 months in either eye
7. Subjects who have had corneal refractive surgery
8. History of Keratoconus, corneal scarring, or other chronic corneal disease in either eye
9. Subjects with contraindication for wearing contact lenses or history of intolerance or difficulties associated with contact lens use including history of dry eye disease
10. Subjects with current signs/symptoms of clinically significant dry eye disease
11. Active eye disease, injury or ocular abnormalities affecting the cornea, conjunctiva, or eyelids or slit lamp findings ≥ grade 3
12. Active inflammation of either eye
13. Active infection of either eye
14. Corneal vascularization of either eye
15. Known allergy to silicone
16. Known allergy to corneal anesthetic
17. Secondary forms of open angle glaucoma (OAG) in either eye
18. Poor or eccentric fixation in either eye
19. Nystagmus
20. Microphthalmos of either eye
21. Buphthalmos of either eye
22. Subject is pregnant, lactating or planning to become pregnant during the course of the study
23. Concurrent participation in any clinical trial
24. Disabling arthritis or limited motor coordination that might limit self-handling of a smart phone with miLens eyepiece attached.
25. Experience using or interacting with miLens and smartphone imaging app during a previous usability or clinical trial
26. Any affiliation with Smartlens and its employees
27. Subjects with any significant dermatologic condition (e.g., history of skin irritation, allergies, skin eczema) that poses a concern for skin contact with the camera eyepiece, based on the Investigator's judgment

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects, aged between 22 and 80 years with:
  1. primary open angle glaucoma (POAG) including normal tension glaucoma
  2. status as POAG suspect including ocular hypertension (OHTN)
  3. no prior diagnosis of POAG/POAG suspect (the subjects in (a) and (b) will henceforth be referred to as "POAG/OHTN" and subjects in (c) will be referred to as "healthy subjects")
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Positive change in miLens output between evening and morning | Through study completion, an average of 1 day
  Positive change in miLens output (via self-operated image acquisition) from evening (the lowest of 6 pm - 7 pm / 7 pm - 8 pm / 8 pm - 9 pm / 9 pm - 10 pm) to morning (the highest of 7 am - 8 am / 8 am - 9 am / 9 am - 10 am / 10 am -11 am)
Repeatability of miLens output using correlation between the Day 0 and Week 1 miLens values | Through study completion, an average of 1 week
  Repeatability of miLens output between Day 0 and Week 1 using correlation between the Day 0 and Week 1 miLens values across the eight time windows (four evening time windows, four morning time windows) for each subject.
Safety of miLens | Through study completion, an average of 1 week
  Frequency and percentage of all ocular and non-ocular adverse events (AE) will be reported. AEs will be categorized by seriousness, relation to device, severity, resolution and use of concomitant medication.

SECONDARY OUTCOMES:
miLens output and iCare correlation | Through study completion, an average of 1 day
  Correlation between iCare measurements (FE) and corresponding miLens measurements.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Nvision Clinical Reseacrh, LLC, Fullerton, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Nvision Clinical Research, LLC, Torrance, California

IPD SHARING:
Plan to Share IPD: No